CLINICAL TRIAL: NCT00790699
Title: A Randomized, Parallel, Single Center, Comparison, Pilot Study Evaluating the Safety and Efficacy of Using Symlin Alongside Insulin in a Multiple Injection Port (I-PORT)
Brief Title: Safety Study of Using Symlin Alongside Insulin in a Multiple Injection Port
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient population
Sponsor: Texas Diabetes & Endocrinology, P.A. (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Thomas C. Blevins, M.D., Thomas Blevins, MD, Texas Diabetes & Endocrinology, P.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDE 001
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: diabetes; Symlin; pramlintide acetate; insulin; multiple injection port; I-PORT
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I-PORT (Active Comparator): Treatment group
  Interventions: Device: I-PORT
- standard injections (Active Comparator): control group
  Interventions: Other: standard injections

INTERVENTIONS:
Device: I-PORT — The study will compare injecting Symlin and insulin into a multiple injection port (I-PORT) vs. standard injections.
  Arms: I-PORT
Other: standard injections — The study will compare injecting Symlin and insulin into a multiple injection port (I-PORT) vs. standard injections.
  Arms: standard injections

SUMMARY:
The purpose of this study is to determine whether injecting Symlin and insulin through a multiple injection port is safe and effective. This will be measured by HbA1c values taken at the beginning of the study and at the final visit.

The secondary objective of the study is to measure patient satisfaction toward using the multiple injection port.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to demonstrate the safety and efficacy of giving pramlintide and insulin in the same multi-port injection device (I-PORT™). Efficacy was measured by HbA1c values taken at baseline and the final visit

The secondary objective of this study is to measure patient satisfaction, opinions and attitudes toward using the I-PORT™ for insulin and pramlintide administration compared to standard insulin and pramlintide injections. The secondary safety and efficacy evaluations included weight, Glycomark, 7-point SMBG evaluations, CGMS evaluations, incidence of glucose values > 300 mg/dl, incidence of glucose values < 70 mg/dl, and insulin dose before the study period, at month 1, 2 and 3.

The primary patient satisfaction evaluations included Quality of Life Questionnaire and treatment satisfaction questionnaires.

The I-PORT™ is a disposable, low profile injection port through which insulin is injected subcutaneously from a standard syringe or insulin pen.(Figure 1) The I-PORT™ allows multiple insulin injections for up to 72 hours. Once the device is applied, the insertion needle is removed and the cannula remains underneath the skin, serving as a delivery channel into the SQ tissue- one skin puncture every three days. To use the device, the subject places the needle on an injection device, such as a syringe or insulin pen, through the re-sealable septum at the top of the I-PORT™ and injects medication directly into the delivery channel.

Study participants included male and females ages 18 and older who were utilizing a regimen of at least two injections daily of rapid acting insulin and at least two injections daily of pramlintide (Symlin®) with an HbA1c between >6.5 and < 9.0%.

There were 39 patients screened for the study and 8 screen failures leaving 31 subjects ages 18 and older, diagnosed with type 1 or type 2 diabetes mellitus for a minimum of six months. 1 patient dropped out of the study due to an AE and 30 completed the study.

A Randomized, Open-Label, Parallel, Single Center, Comparison Study. Approximately 13 patients with type 1 diabetes and 18 patients with type 2 diabetes were randomized into one of two treatment groups. The randomization was stratified within diabetes type (1 vs. 2) and low (6.5-7.5) vs. high (7.6-9.0) HbA1c level. The randomization process was executed using a computer generated randomization table.

Subject Groups:

* Group 1- Study subjects administered insulin and pramlintide using standard injection therapy during the entire duration of the trial
* Group 2- Study subjects administered insulin and pramlintide via a single I-PORT™ for the entire duration of the trial

This study consisted of 8 visits: Screening/Visit 1, Visit 1a (Day -3), Visit 2 (Baseline/Day 0), Visit 3(Day 14), Visit 4(Month 1), Visit 5(Month 2), Visit 5a (Day 81) Visit 6(Month 3).

Subjects participating in this protocol were asked to take their rapid acting insulin preparations and Pramlintide (Symlin®) at the same time using the dose called for by their prescribed regimen established prior to study entry. Subjects used their usual type of insulin preparations obtained by prescription from the commercial pharmacy system. Subjects randomized into Group 2 were given guided instruction on the proper technique of insertion, use and removal of the I-PORT™.

I-PORT™ devices were provided to the subjects and dispensed throughout the trial. Pramlintide (Symlin) was supplied by Amylin Pharmaceuticals.

Patients performed a 7 point SMBG test 3-5 days at baseline and all subjects were instructed on use of a Continuous Glucose Monitoring System (Medtronic iPro). The sensor was inserted for 3-day wear at baseline and blood samples for HbA1c and Glycomark testing were obtained. All subjects completed treatment satisfaction and QoL questionnaires. Each subject was randomized to one of two possible treatment groups.

At each visit, subject diaries were reviewed, weight measurement and a site insertion exam were performed. AEs and concomitant medications were reviewed at each visit.

Patients were asked to do a 7 point SMBG test 3-5 days prior to visit 3,4,5, and 5a. At visit 5a subjects were again instructed on use of a CGMS and a sensor was inserted for 3-day wear.

At the final visit (visit 6), the CGMS was removed and treatment satisfaction and QoL questionnaires were completed by all subjects, and blood samples were taken for HbA1c and Glycomark testing.

Patients were instructed to contact the site if they had 2 glucoses in a row > 300 mg/dl or 2 glucoses in a row of <70 mg/dl. Insulin and/or Pramlintide (Symlin®) were adjusted by PI as needed throughout the trial. Discontinuation of I-PORT™ use was at the discretion of the PI as a rescue measure.

The following QoL questionnaires/ Treatment satisfaction questionnaires were obtained from patients at screening and at the final visit: DSTQ, DSTQ-c, DDS, TSQ,I-PORT™ Device Benefits, Insulin/Symlin Satisfaction Questionnaire, I-PORT™ Device Management, General Diabetes Management, I-PORT™ Device Satisfaction

ELIGIBILITY:
Inclusion Criteria:

* male or female ages 18 and up
* utilizing a regimen of at least two injections daily of insulin and at least two injections daily of Symlin
* able to understand and sign an informed consent form and HIPPA form
* agrees to all study visits and procedures
* HbA1c between >6.5 and <9.0 (inclusive)

Exclusion Criteria:

* history or current diagnosis of chronic disease which in the view of the PI would interfere with adequate involvement in and completion of the requirements of the study
* history of malignancy with in the last five years of study entry (other than basal cell carcinoma)
* current use of any drugs that alter gastrointestinal motility (e.g., anticholinergic agents such as atropine), agents that slow intestinal absorption of nutrients (e.g. a-glucosidase inhibitors) or promotility agents (e.g. metaclopromide)
* any contraindication of Symlin or I-PORT according to the package labeling
* are female and pregnant, lactating or planning to become pregnant during the duration of the trial
* are poorly compliant with their current insulin and/or Symlin regimen, as defined by their HCP
* has history of known hypersensitivity to plastics or polymers
* treatment with any investigational drug within one month prior to enrollment
* myocardial infarction or stroke within six months prior to screening
* initiated use of Symlin pen or any Insulin pen in lieu of a vial in last 4 weeks (pen use is okay as long as they have been using it for at least 4 weeks prior to screening visit)
* female subjects of childbearing potential practicing inadequate birth control (adequate birth control is defined as using oral contraceptives, double barrier methods, Intrauterine devices, surgical sterilization or vasectomized partner)
* have confirmed diagnosis of gastroparesis
* have hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Blevins, MD, Principal Investigator — Texas Diabetes & Endocrinology
Locations (1):
- Texas Diabetes & Endocrinology, PA, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Injections: standard injections: The study will compare injecting Symlin and insulin into a multiple injection port (I-PORT) vs. standard injections. The standard injections are usually 3-4 times daily.
Period: Overall Study
Arm/Group | I-PORT | Standard Injections
Started | 17 | 14
Completed | 16 | 14
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I-PORT | Standard Injections | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (16.38) | 54 (10.60) | 49.5 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 15 | 10 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 31
Glycomark [Mean (Standard Deviation); unit: ug/mL] | 6.49 (3.69) | 5.05 (3.71) | 5.84 (3.71)
Type of Diabetes Breakdown [Count of Participants; unit: Participants]
  Type 1 Diabetics | 7 | 6 | 13
  Type 2 Diabetes | 10 | 8 | 18
Type 1 diabetes [Count of Participants; unit: Participants] | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be Measured by HbA1c Values Taken at Screening, Baseline and After Three Months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | I-PORT | Standard Injections
Number analyzed (Participants) | 17 | 14
% of HbA1c
  Screening | 7.68 (.65) | 7.93 (.73)
  Month 3 | 7.34 (.60) | 7.42 (.90)
  Baseline | 7.66 (.35) | 7.70 (.67)

2. Secondary Outcome: The Secondary Outcome Will Measure Patient Satisfaction, Opinions and Attitudes Toward Using the Multiple Injection Port for Insulin and Symlin Administration Compared to Standard Symlin Injections (Measured Through Using Questionnaires).
Description: Scores from the QOL and treatment satisfaction measures collected at Visit 1 and Visit 6.
  To determine if patient satisfaction and patient opinions and attitudes toward using the I-PORT™ for insulin and Symlin® administration compared to standard insulin and Symlin® injections was significantly different for patients in the treatment and control groups, repeated-measures analysis of variance (RM-ANOVA) was conducted on scores from the quality of life and treatment satisfaction measures collected at Visit 1 and Visit 6. The RM-ANOVA results were evaluated to determine if any statistically significant changes occurred. TSQ- lower numbers show less satisfied. DDS- Lower numbers show decrease in distress. DTSQ- Lower numbers show less satisfied. One patient did not complete Visit 6 questionnaires.
  Scale ranges:
  DDS scale range: 17- 102 DTSQc scale range: 16- 96 Insulin /Symlin Treatment Satisfaction Questionnaire scale range: 15-90
Time Frame: 3 months
Population: Results broken down further to reflect results in each group: Iport vs. Standard Injection subjects and total number of subjects who completed the patient reports at visit 1 and Visit 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Visit 1: Patient reports at visit 1
- Visit 6: Patient reports at last visit (3 months)
Arm/Group | Visit 1 | Visit 6
Number analyzed (Participants) | 31 | 30
units on a scale
  Treatment Satisfaction Control: number analyzed (Participants) | 14 | 14
  Treatment Satisfaction Control | 66.07 (13.34) | 65.66 (13.94)
  Treatment Satisfaction Treatment: number analyzed (Participants) | 17 | 16
  Treatment Satisfaction Treatment | 67.16 (12.30) | 54.28 (16.71)
  DTSQ Control: number analyzed (Participants) | 14 | 14
  DTSQ Control | 37.46 (5.95) | 34.54 (7.40)
  DTSQ Treatment: number analyzed (Participants) | 17 | 16
  DTSQ Treatment | 35.41 (6.78) | 33.25 (6.15)
  Diabetes Distress Scale Control: number analyzed (Participants) | 14 | 14
  Diabetes Distress Scale Control | 38.20 (10.56) | 33.86 (8.19)
  Diabetes Distress Scale Treatment: number analyzed (Participants) | 17 | 16
  Diabetes Distress Scale Treatment | 34.00 (10.57) | 31.45 (10.74)
Statistical Analysis 1: Comparison: Visit 1 vs Visit 6; The results were evaluated to determine if any statistically significant changes in any of these measures between the first and final visit occurred and if these changes were associated with membership in the treatment or control group; Test type: Superiority or Other; p > .05, RM-ANOVA

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Iport: Treatment group/ Iport Users
- Standard Injections: Control group/ Standard Injections
Arm/Group | Iport | Standard Injections
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 11/16 | 7/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iport (N=16) | Standard Injections (N=14)
Upper respiratory infections (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infections (Infections and infestations) | 2 (2) | 0 (0)
Common Cold (Infections and infestations) | 1 (1) | 2 (2)
uterine ablation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperglycmia (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
left wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dental implants (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Yeast infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parvo Virus (Infections and infestations) | 1 (1) | 0 (0)
Trigger finger release (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mettalic taste (General disorders) | 1 (1) | 0 (0)
mettalic smell (General disorders) | 1 (1) | 0 (0)
confusion (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Black liquid stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Boil (General disorders) | 0 (0) | 1 (1)
swollen lymph node (General disorders) | 0 (0) | 1 (1)
dizziness (General disorders) | 0 (0) | 1 (1)
tooth abcess (Infections and infestations) | 0 (0) | 1 (1)
bacterial bronchitis (Infections and infestations) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No